CLINICAL TRIAL: NCT00785993
Title: Impact of Egg-Banking in an Ovum-donation Program
Brief Title: Egg-Banking and Ovo-donation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Ana Cobo, Instituto Valenciano de Infertilidad, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0703-C-017-AC
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Egg Banking
Keywords: Egg banking, clinical outcome

ARMS (2):
- Control Group (Active Comparator): Fresh donor oocytes
  Interventions: Other: Protocolary IVF treatment with fresh donor oocytes
- Group I (Experimental): vitrified donor oocytes
  Interventions: Other: Vitrification of oocytes for IVF treatment

INTERVENTIONS:
Other: Vitrification of oocytes for IVF treatment
  Arms: Group I
Other: Protocolary IVF treatment with fresh donor oocytes
  Arms: Control Group

SUMMARY:
Egg-banking would considerably simplify the logistics and means by which oocytes could be donated. These banks would make it easier to immediately provide oocytes that would be compatible to the recipient, shortening or even eliminating the problem of long waiting lists. Egg-banking would also allow the oocytes to be effectively quarantined, drastically diminishing the risk of transmission of infectious diseases in a fashion analogous to semen banks. The most essential prerequisite for a successful egg cryo-banking program is to have an efficient oocyte cryopreservation technology. Recent studies, including our own experience, have indicated that vitrified oocytes preserve intact their potential to fertilize and further develop into competent embryos, giving high clinical results as well as high survival rates. The aim of this study is to evaluate impact of the establishment of an egg-banking in our ovum donation program. Oocyte cryopreservation is carried out by Cryotop method. The study includes oocyte donation cycles conducted with fresh and vitrified oocytes. Recipients are allocated randomly into each group ("fresh vs. vitrified cycles"). Main outcome measures include survival, fertilization, embryo development and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Receptors

  * Women receiving donor oocytes and whose partners without seere pathology of semen.
  * BMI < 25

Donors:

Inclusion Criteria:

18 - 35 years oldaños.

* Normal Response (8-15 follicles)to long protocol of ovarian stimulation with hCG
* Donors with normal menstrual cycles ( 21-35 day duration).
* Donors with Body Mass Index (BMI) between 18-25 Kg/m2

Exclusion Criteria:

* Donors with +/= two previous miscarriages'
* Polycystic Ovary Syndrome
* Donors with antecedents of poor embrionary quality not attributed to masculine factor.
* Donors with decline of Estradiol Hormone of more than 10% or Estradiol Hormone plateau.
* Donors with a high response >20 ovocitos and/or levels above 3000pg/mL of Estradiol the day of the administration of Chorionic gonadotropin (hCG.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical outcome in an ovum donation program conducted with egg-banking. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cobo, PhD, Principal Investigator — Instituto Valenciano de Infertilidad
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Cobo A, Meseguer M, Remohi J, Pellicer A. Use of cryo-banked oocytes in an ovum donation programme: a prospective, randomized, controlled, clinical trial. Hum Reprod. 2010 Sep;25(9):2239-46. doi: 10.1093/humrep/deq146. Epub 2010 Jun 30. PMID 20591872